CLINICAL TRIAL: NCT06505668
Title: Effect Of Atenolol Versus Ivabradine On Heart Rate Variability In Treatment Resistant Schizophrenia Patients On Clozapine With Tachycardia: A Randomized Control Trial.
Brief Title: Effect of Atenolol Versus Ivabradine on HRV in TRS Patients on Clozapine With Tachycardia: A Randomised Control Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Professor and Head, Department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIIMSBBSR/PGThesis/2023-24/90
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Treatment Resistant Schizophrenia; Clozapine Adverse Reaction; Heart Rate Variability; Tachycardia
Keywords: Clozapine; Treatment resistant schizophrenia; heart rate variability
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Tachycardia | interventions — Atenolol; Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atenolol 25mg (Active Comparator): Patients will be receiving Atenolol 25mg OD for 2 months.
  Interventions: Drug: Atenolol 25 mg
- Ivabradine 10mg (Active Comparator): Patients will be receiving Ivabradine 10mg (5mg BD) for 2 months.
  Interventions: Drug: Ivabradine 10mg

INTERVENTIONS:
Drug: Atenolol 25 mg — Patients will be receiving Atenolol 25mg OD for 2 months.
  Other Names: Arm A
  Arms: Atenolol 25mg
Drug: Ivabradine 10mg — Patients will be receiving Ivabradine 5mg BD for 2 months.
  Other Names: Arm B
  Arms: Ivabradine 10mg

SUMMARY:
Clozapine is the only drug approved for Treatment Resistant Schizophrenia. However, it has been associated with many adverse drug reactions including agranulocytosis, myocarditis, sialorrhea, constipation, orthostasis, tachycardia. There are many factors that have impacted the use of clozapine in TRS patients including physician hesitation, patient denial, stopping of drug due to Adverse drug reactions.

Although Tachycardia should not be the reason to stop clozapine, but data shows that it leads to discontinuation of drugs in significant patient population. If patient on clozapine develops tachycardia; first orthostasis, myocarditis and systemic infection should be ruled out. Tachycardia traditionally have been treated with B1 adrenergic blockers such as Atenolol. But the problem with beta blocker medications is that significant proportion develops hypotension.

Recently developed Ivabradine slows heart rate via I(f) current, and is not associated with much cardiac adverse effects. Recent Clinical trials have been carried out to show its effects on Clozapine associated tachycardia which shows promising results. Some studies suggest using Ivabradine in patient population that have contraindication for beta blockers.

Although both of these drugs are used widely in clinical practice, but as Ivabradine is relatively new drug there have been no head-to-head comparison with Atenolol. A recent meta-analysis tried to compare treatment efficacy in these patients, but found no studies that met their inclusion criteria. This current study attempts to make such comparison and guide further research.

DETAILED DESCRIPTION:
Schizophrenia is a severe debilitating mental disorder characterised by distortions of thinking, perception and blunt affect. It poses a major healthcare burden with the prevalence of 1% worldwide. As per National Mental Health Survey of India (2016), the prevalence of Schizophrenia and other psychotic disorders was 0.4% and the lifetime prevalence was 1.4%. The earliest success in treating some of the symptoms of schizophrenia came with the discovery of typical antipsychotics. Later, newer "atypical" antipsychotics with different psychopharmacological actions promised better outcomes, but were found similar in clinical response although with less extrapyramidal side effects.

Almost 30% patients with schizophrenia do not show clinically significant improvement with antipsychotic medications. Treatment resistant schizophrenia (TRS) is thus, defined as inadequate response to at least two failed antipsychotic trials of adequate dose and duration. However, clozapine has been found to be exceptionally effective in such cases.

Therefore, multiple guidelines including FDA approve clozapine as the only pharmacological agent in the treatment for TRS. However, its use is associated with serious myocarditis, agranulocytosis, seizures and sudden cardiac death along with a plethora of common side effects like sedation, weight gain, constipation, hypersalivation, tachycardia, orthostatic hypotension. Clozapine causes dysregulation of the autonomic nervous system possibly by anti-muscarinic effects and inhibition of vagal neurons resulting in constipation, orthostasis, tachycardia. The side-effects of clozapine has been notoriously the major cause behind its underutilisation under clinical settings, therapeutic challenge due to need for constant monitoring of the physical and blood parameters of the patients and high rates of treatment dropouts. For instance, persistent tachycardia occurs in approximately 33% of TRS receiving clozapine ultimately leading to treatment discontinuation in at least 10% of cases. Moreover, high heart rate has been an independent predictor for cardiovascular diseases, stroke, sudden cardiac death and noncardiac diseases. It has been shown that for each rise in 10 bpm from resting heart rate the relative risk for these diseases increases linearly. Therefore, there is a need to understand the effects of clozapine on the autonomic nervous system, and regularly monitor the relevant parameters for early detection and intervention to ensure treatment adherence, prevention of any serious cardiac event and improve the overall quality of life of these patients.

One way to measure autonomic dysregulation induced by clozapine is with the help of heart rate variability. Heart Rate Variability (HRV) is the change in time duration of adjacent heart beats, arising from various mechanisms including but not limited to brain-heart interaction, blood pressure, gaseous exchange, vascular tone, hormone levels. HRV can be measured in different time periods (ultra-short-term(<5min), short-term (5min) and 24hours measurement)and described into different metrics (including time-domain, frequency-domain and non-linear measurements). The time-domain includes interbeat duration variation as measured by standard deviation of all interbeat duration, root mean square of all interbeat duration etc. Frequency-domain is analysed using Power spectral density (PSD) calculated using Fast Fourier Transformation (FFT) . When measuring for short-term, frequency-domain should be preferred. Due to its antimuscarinic effects, Clozapine has shown to cause high mean heart rate, low heart rate variability, high low-frequency component when compared to other antipsychotics or control patients.

Most guidelines suggest treating persistent tachycardia in patients receiving clozapine after excluding other causes of tachycardia. Beta blockers (like Atenolol) or Calcium channel blockers have been recommended for clozapine associated tachycardia (20). Patients who do not tolerate these drugs can be prescribed Ivabradine. The exact mechanism by which Ivabradine modulates autonomic function is not known, but is hypothesised to be its effects on the intra cardiac nervous system, which by a feedback to the Central Nervous System via the afferent nerve fibres from the heart results in overall increase in the parasympathetic activity.

The available literature is scarce about the effects of clozapine on the heart rate variability. Moreover, despite the usual prescription of beta blockers/ ivabradine in the treatment of the clozapine induced tachycardia, evidence for the same are limited in the specific population of TRS patients. Furthermore, all studies supporting their use has been conducted in western countries. Again, there is no clear consensus regarding the choice of one drug over the other, given their different pharmacodynamic actions. The specific effects of these drugs (beta blockers/ ivabradine) on the HRV caused by clozapine therefore needs further exploration. This study is intended to compare the effects of atenolol versus ivabradine on heart rate variability in patients of TRS on Clozapine with tachycardia. The findings of the study will be able to guide appropriate use of the mentioned pharmacological therapies in context of clozapine-induced autonomic instability/tachycardia. This will help improve the overall cardiac functioning and the tolerability and compliance in TRS scenarios.

ELIGIBILITY:
Inclusion Criteria:

All patients coming for treatment at the Out-patient department and In-patient department of the Department of Psychiatry fulfilling the following are included:

1. Patients diagnosed with TRS (TRRIP consensus) receiving clozapine.
2. Aged between 18 to 60 years of either sex
3. Having baseline heart rate of >100/minute.
4. Written informed consent from Legally Authorized representative.

Exclusion Criteria:

Patients with any one of the following are excluded from the study:

1. Already receiving Atenolol or Ivabradine.
2. Patients having any contraindication to using Atenolol or Ivabradine.
3. Receiving any other medication other than Clozapine known to cause autonomic dysregulation.
4. Active substance use.
5. Serious medical or neurological comorbidity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of Atenolol vs Ivabradine as changes in the Frequency domain of HRV over 2 months. | 2 months
  Change in frequency domain parameters of participants will be compared between both the arms.

SECONDARY OUTCOMES:
To compare the changes in the time domain of HRV between the groups. | 2 months
  Change in the time domain parameters of participants will be compared between both the arms.
To compare the changes in central & peripheral BP and Pulse Rate between the groups. | 2 months
  Change in the time domain parameters of participants will be compared between both the arms.
To find any correlation between the severity of PANSS with HRV at baseline. | single measure
  PANSS will be applied at the baseline and will be correlated with HRV parameters of all participants.
To compare the treatment emergent adverse reaction over 2 months between the groups. | 2 months
  All the participants will be kept in contact throughout the intervention period and will be screened for any adverse drug reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Biswa Ranjan Mishra, MD, Principal Investigator — Professor and Head, Department of Psychiatry
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
It will be decided later on.